CLINICAL TRIAL: NCT01558804
Title: Gene Expression in Isolates of Group A Streptococci Recovered From Patients Who Are Carriers
Brief Title: GRoup A StrePtococcus
Acronym: GRASP
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2011-0058; 2015-1456 (Other: Institutional Review Board - 5 year replacement); A536700 (Other: UW Madison); SMPH\PEDIATRICS\PEDIATRICS (Other: UW Madison); 1R21AI147502-01 (NIH); Protocol Version 9/14/2023 (Other: UW Madison)
Record Dates: First submitted 2012-03-08; First posted 2012-03-20 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Streptococcal Pharyngitis
Keywords: Streptococcus pyogenes; Streptococcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Throat swab specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rapid Strep Positive: Children will be eligible for this study if they are ages 5 to 15 years and have been diagnosed to have acute pharyngitis caused by GAS with a positive Rapid Antigen Detection Test (RADT).
  Interventions: Other: Identifying group A strep carriers

INTERVENTIONS:
Other: Identifying group A strep carriers — At study entry, at 14 days, and if follow up is positive, again in 14-21 days: Standard culture for GAS and analysis of mRNA.

SUMMARY:
The purpose of the research is to help understand why some children become carriers of strep and whether children who are carriers need to be treated with antibiotics.

DETAILED DESCRIPTION:
The overall objective of this investigation is to understand the differences in Group A streptococci in children who are acutely infected from those who are carriers. The hypothesis is that when in the carrier state, GAS exhibits unique transcriptional profiles that differ from those of the acute infection state. The investigators expect transcriptional profiles of GAS to provide important information regarding the changes the organism undergoes when transitioning between acute infection and carriage.

The specific aims of this study are:

1. To collect longitudinal participant-samples from acute and carriage phases of GAS infection and compare transcriptomic profiles and whole genome sequences of GAS recovered from acute and carrier pharyngeal swabs obtained from the same participants.
2. To evaluate how identified differentially expressed genes, or observed genetic polymorphisms, influence GAS models of bacterial colonization and pathogenesis.

To do this, the investigators will to identify 12 children with acute pharyngitis due to Group A streptococcus (GAS) who are pharyngeal carriers of GAS. Thirty percent of children 4 to 16 years of age with acute pharyngitis occurring between October and May will have a positive culture or rapid antigen detection test for GAS. Approximately 8-10% of these children with pharyngitis and a positive culture or rapid antigen detection test (RADT) for GAS will be carriers. Therefore,180 participants will need to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 5-15 years
* Positive rapid antigen detection test for group A streptococcus
* Parent or legal guardian present and able to provide consent
* Provider prescribes treatment with a beta lactam antibiotic
* English speaking

Exclusion Criteria:

* Unable to take beta lactam antibiotics
* Other concurrent bacterial infection, i.e., pneumonia

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be eligible for this study if they are ages 5 to 15 years and have been diagnosed to have acute pharyngitis caused by GAS (with a positive rapid antigen detection test (RADT). Children will be excluded if they are unable to take beta lactam antibiotics. Children will be enrolled at UW Health sites in Madison, Wisconsin, including both pediatric ambulatory care clinics and urgent care clinics. The study team will offer participants the option to complete follow-up study visits in-clinic
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2011-05-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Identifying children who are pharyngeal carriers of Group A streptococcus | 2 weeks
  The specific aim of this study is to identify 30 children with acute pharyngitis due to Group A streptococcus (GAS) and 30 children who are pharyngeal carriers of GAS.
  Thirty percent of children 4 to 16 years of age with acute pharyngitis occurring between October and May will have a positive culture or rapid antigen detection test for GAS. Approximately 10-15% of these children with pharyngitis and a positive culture or rapid antigen detection test (RADT) for GAS will be carriers

CONTACTS AND LOCATIONS:
Overall Officials: Gregory DeMuri, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health Pediatric Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisno AL. Acute pharyngitis. N Engl J Med. 2001 Jan 18;344(3):205-11. doi: 10.1056/NEJM200101183440308. PMID 11172144
- [Background] Carapetis JR, Steer AC, Mulholland EK, Weber M. The global burden of group A streptococcal diseases. Lancet Infect Dis. 2005 Nov;5(11):685-94. doi: 10.1016/S1473-3099(05)70267-X. PMID 16253886
- [Background] Musser JM, Shelburne SA 3rd. A decade of molecular pathogenomic analysis of group A Streptococcus. J Clin Invest. 2009 Sep;119(9):2455-63. doi: 10.1172/JCI38095. PMID 19729843
- [Background] Pichichero ME. Group A beta-hemolytic streptococcal infections. Pediatr Rev. 1998 Sep;19(9):291-302. doi: 10.1542/pir.19-9-291. PMID 9745311
- [Background] Jiang H, Wong WH. Statistical inferences for isoform expression in RNA-Seq. Bioinformatics. 2009 Apr 15;25(8):1026-32. doi: 10.1093/bioinformatics/btp113. Epub 2009 Feb 25. PMID 19244387
- [Background] Li J, Jiang H, Wong WH. Modeling non-uniformity in short-read rates in RNA-Seq data. Genome Biol. 2010;11(5):R50. doi: 10.1186/gb-2010-11-5-r50. Epub 2010 May 11. PMID 20459815
- [Background] Anders S, Huber W. Differential expression analysis for sequence count data. Genome Biol. 2010;11(10):R106. doi: 10.1186/gb-2010-11-10-r106. Epub 2010 Oct 27. PMID 20979621
- See also: University of Wisconsin-Madison Department of Pediatrics Research Information — http://www.pediatrics.wisc.edu/research/